CLINICAL TRIAL: NCT02480660
Title: Adolescent to Adult-Oriented Health Care Transition Survey: Study of a Video-Based Educational Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: Academic Pediatric Association (Industry)
Responsible Party: Principal Investigator, Keely Dwyer-Matzky, Assistant Professor, University of Rochester
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: RSRB00044255
Record Dates: First submitted 2015-05-01; First posted 2015-06-24 (Estimated); Last update posted 2016-02-22 (Estimated); Status verified 2015-06

CONDITIONS: Transition to Adult Health Care
Keywords: Hospitalized; adolescents; knowledge; transition; educational intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Video Intervention Group (Experimental): Subjects will be randomized to intervention group where participants will be asked to watch a 7 minute educational video.
  Interventions: Behavioral: Educational Video
- Control Group (No Intervention): Subjects will be randomized to control group ( no intervention) and receive standard of educational care on adolescent to adult oriented health care transitions.

INTERVENTIONS:
Behavioral: Educational Video — The video highlights key elements found in the existing literature critical for transition including understanding and taking charge of their health, creating a medical summary, learning more about health insurance, introducing the idea of organizing a health care transition team and creating a plan. The video also educates patients on the opportunities to take a tour of an adult floor, talk with social workers and learn more about adult providers during their hospital stay.
  Arms: Video Intervention Group

SUMMARY:
Purpose: To understand the baseline knowledge on the transition of care to adult providers in hospitalized adolescent patients and to test if an educational intervention given during an inpatient stay in a medium size academic pediatric hospital affects perception of knowledge, attitudes and participation in transition planning.

Primary Research Question: Will a video-based educational intervention in an academic pediatric hospital affect perception of knowledge, attitudes and participation in transition planning to adult oriented health care of the hospitalized adolescent?

Secondary Research Question: What is the baseline experience of the hospitalized adolescent in key elements of transitioning to adult oriented health care?

DETAILED DESCRIPTION:
Purpose: To understand the baseline knowledge on the transition of care to adult providers in hospitalized adolescent patients and to test if an educational intervention given during an inpatient stay in a medium size academic pediatric hospital affects perception of knowledge, attitudes and participation in transition planning.

Aim 1: To determine the effect of viewing a video-based educational intervention in an academic pediatric hospital affect perception of knowledge, attitudes and participation in transition planning to adult oriented health care of the hospitalized adolescent.

Aim 2: To describe the baseline experience and knowledge base of hospitalized adolescents regarding key elements of transitioning to adult-oriented health care.

CHARACTERISTICS OF THE RESEARCH POPULATION

1. Number of subjects: There will be approximately 140 subjects assuming approximately 50% attrition by the third survey.
2. Gender of Subjects: Subjects of either gender will be part of the study. Discrepancies in gender will be related to the patient population at the time of the study enrollment.
3. Age of Subjects: The age range will be 15 to 25 years old.
4. Racial and Ethnic Origin: There will be no enrollment restrictions based on race. It is expected that the racial distribution of our study population will mirror that of the inpatient pediatric patient population.

Methods and Procedures:

The purpose of the study will be achieved by surveying all eligible subjects admitted to the children's hospital. Eligible patients will be identified by the daily unit census in the children's hospital, excluding the patients outlined under exclusion criteria. Informed consent will be obtained from their parents and patients will assent to participate in the study. Personal health information and contact information will be collected with parents present by study investigator prior to randomization of subjects and will be stored separately from other survey data stored in a secure database on a password protected computer. All paper files will be kept in a locked office.

1. At the time of enrollment patients will be stratified by age for block randomization in order to have balanced intervention and control groups. The age groups will be 15-16 year old control or intervention group vs 17 years old and greater control or intervention group. Both groups will be asked to complete three surveys during the course of the study; in terms of education, the control groups will receive standard care education while the intervention group will view an educational video on transition from adolescent to adult oriented health care. All subjects will be oriented to the use of the Get Well Network in order to access the surveys via SurveyMonkey© (Palo Alto, CA). The first survey will consist of 40 questions. A number of first survey questions were obtained and modified from the web questionnaire of 2007 Survey of Adult Transition and Health (SATH) from Department of Health and Human Services, Maternal and Child Health Bureau (MCHB) of the Health Resources and Services Administration (HRSA). Other questions from the Health-Care, Self Determination questionnaire packets relating to treatment self-regulation and perceived competence have been modified to focus on independence in health care management.
2. After completing the first survey the intervention group subject will then be prompted via an embedded html link within the survey to watch a seven minute educational video.
3. Prior to discharge from the hospital, participants in both groups will be asked to complete a second survey assessing willingness to prepare for the transition to adult oriented medical care, and actions taken during the hospital stay. Possible actions include taking a tour of an adult unit, discussing health insurance changes with a social worker, asking for a copy of a sample medical summary or requesting information about adult primary care and/or specialty providers. Patients will be given a reminder in person or via Facebook, phone, text or e-mail to complete the second survey via SurveyMonkey.
4. Approximately 4 weeks after hospital discharge a reminder via Facebook, phone, text or e-mail will be sent to complete the third survey via SurveyMonkey©. If the subject does not have access to the internet, then the survey will be administered by phone.

A retrospective chart review will be performed to record each subject's type of health insurance and chronic illness based on the medical chart from the current hospitalization. Comparison will be made between the patient's awareness of his underlying chronic illness and compared with health care providers' documentation of underlying chronic illness.

Data Analysis and Monitoring Data will be statistically analyzed using descriptive statistics such as mean and standard deviation, chi square testing and regression analysis. Excel, SPSS and SAS will be used for statistical calculations. Dr. Keely Dwyer-Matzky , the principal investigator will be responsible for ensuring the privacy of the data. Since there is minimal risk a data and safety monitoring plan is not necessary.

Data Storage and Confidentiality

SurveyMonkey© is a confidential proprietary survey tool that collates quantitative data and written comments into convenient reports. SurveyMonkey© uses Secure Sockets Layer (SSL) technology, which protects user information through both server authentication and data encryption, ensuring that user data is safe, secure, and available only to authorized persons. Investigators will protect all health identifiers. Data downloaded from SurveyMonkey© will be maintained on electronic files on a secure server with password protection. Only authorized researchers will have access to the data. University of Rochester Office of Human Subjects or research regulatory groups may review these records.

ELIGIBILITY:
Inclusion Criteria:

* All subjects admitted to Golisano Children's Hospital from 15 to 25 years old except those defined by exclusion criteria

Exclusion Criteria:

* Critically ill, as defined as being ICU patients;
* Patients with acute psychosis;
* Patients boarding within the pediatric hospital admitted to an adult hospital service;
* Patients who have previously viewed the video;
* Intellectually disabled;
* Non -English speaking subjects and patients who have previously participated in the study.
* For patients with an intellectual disability investigators will defer to the parents' judgment whether the patient can complete the surveys independently.

Ages: 15 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 152 (Actual)
Dates: Start 2013-11; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Measure the number of subjects who showed a positive change in perception of transition knowledge in survey responses pre and post intervention | 2 years
  Will measure primary outcomes using likert scales ( eg very interested, somewhat interested, not very interested and not interested) Will compare pre and post intervention in intervention group and will compare intervention group to control group pre and post intervention.
Measure the number of subjects who showed a positive change in attitudes about transition in survey responses pre and post intervention. | 2 years
  Will measure primary outcomes using likert scales ( eg very interested, somewhat interested, not very interested and not interested) Will compare pre and post intervention in intervention group and will compare intervention group to control group pre and post intervention.
Measure the number of subjects who showed a positive change in participation in transition planning in survey responses pre and post intervention | 2 years
  Will measure primary outcomes using likert scales ( eg very interested, somewhat interested, not very interested and not interested) Will compare pre and post intervention in intervention group and will compare intervention group to control group pre and post intervention.

SECONDARY OUTCOMES:
Measure the number of subjects who had a positive baseline survey response in hospital experience | 2 years
  Will measure secondary outcome measures using likert scales ( eg very interested, somewhat interested, not very interested and not interested) Will compare all respondents based on age, race, gender, special health care need, health insurance and education level.

CONTACTS AND LOCATIONS:
Overall Officials: Keely E Dwyer-Matzky, MD, Principal Investigator — University of Rochester
Locations (1):
- Golisano Children's Hospital at Strong, Rochester, New York, United States